CLINICAL TRIAL: NCT04915521
Title: Effect of Ultrasound-guided Erector Spinalis Plane Block on Postoperative Pain and Intraoperative Opioid Consumption in Bariatric Surgery
Brief Title: Erector Spinalis Plane Block in Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meliha Orhon (Other)
Responsible Party: Sponsor-Investigator, Meliha Orhon, assistant professor, Marmara University
Organization: Marmara University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 09.2020.128
Record Dates: First submitted 2021-04-19; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Postoperative Pain; Opioid Consumption
Keywords: bariatric surgery; morbid obesity; ultrasound-guidance; erector spinalis plane block (ESPB); visual analogue scale (VAS) score; opioids
MeSH Terms: conditions — Pain, Postoperative; Obesity, Morbid | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- erector spinae plane block group (Active Comparator): ESPB group received ultrasound-guided bupivacaine and lidocaine injection at T9 vertebral level before anesthesia induction.
  Interventions: Other: erector spina plane block (ESPB) group
- non block control group (No Intervention): Control group received 5 ml 0.5% bupivacaine injection to each trocar site (total of 25 ml) at the beginning of the operation.

INTERVENTIONS:
Other: erector spina plane block (ESPB) group — An experienced anesthesiologist performed ESPB in all patients in sitting position bilaterally.
  A linear ultrasound probe (6-13 MHz) was used for ultrasound guidance. Injection was done using in-plane technique. A 22G block needle (100mm, B-Braun, Germany) was inserted 3- cm lateral to the T9 spinous process and advanced in cranio-caudal direction. To separate erector spina muscle from the transverse process, initially 1-2 ml saline was injected; then 20 ml 0.5% bupivacaine and 5 ml 0.2% lidocaine were injected following separation. Diffusion of the drugs in erector spina plane at cranio-caudal line was ensured. No analgesic or sedative was used during the procedure.
  Other Names: non-block control group
  Arms: erector spinae plane block group

SUMMARY:
Background/objective: Bariatric surgery is often associated with moderate to severe pain. In obese individuals, opioids have the potential to induce ventilatory impairment; thus, opioid use needs to be limited. This study aimed to compare the novel ultrasound-guided erector spinalis plane block (ESPB) technique with controls in terms of intraoperative opioid consumption and postoperative pain control. Methods: A total of 63 patients with morbid obesity who underwent laparoscopic bariatric surgery were included in this randomized study. Patients were randomly assigned to the bilateral erector spina plane block (ESPB) group or the control group. To evaluate perioperative pain and to adjust opioid dose, analgesia nociception index (ANI) was monitored during surgery. Total opioid dose was recorded for each patient. In addition, pain was evaluated using visual analogue scale (VAS) scores for 24 hours following the operation.

DETAILED DESCRIPTION:
Obesity represents a major disease burden and healthcare challenge globally due to its increasing prevalence over the last decades. From 1980 to 2013, worldwide prevalence of overweight/obesity increased by 27·5% for adults and 47·1% for children, resulting in an estimated global total number of obese/overweight individuals slightly more than two billion. Obesity is associated with serious conditions including cardiovascular disease, diabetes, some cancers, kidney disease, sleep apnea, gout, osteoarthritis, hepatobiliary disease, resulting in increased mortality and decreased life expectancy among obese individuals. On the other hand, weight loss leads to improvement of these conditions and outcomes. Life-style modifications with diet, exercise, and behavioral therapy, pharmacotherapy, and surgery are used for the management of obesity. Bariatric surgery represents an effective and a sustainable treatment modality in patients with morbid obesity, laparoscopic sleeve gastrectomy and gastric bypass being the most common procedures. However, these procedures are mostly associated with moderate to severe postoperative pain, which is often a combination of abdominal wall pain and visceral pain.Postoperative pain, when not adequately controlled, has unfavorable consequences such as impaired quality of life and recovery as well as increased risk of surgical complications and persistent postsurgical pain. Patients with morbid obesity represent a special group when it comes to perioperative pain management. These patients have a higher incidence of sleep-disordered breathing; therefore, opioids have the potential to induce ventilatory impairment resulting in increased morbidity/mortality. Stepwise and severity based-multi-modal analgesia with opioid-sparing approach can improve safety; thus, Enhanced Recovery After Surgery (ERAS) guidelines for bariatric surgery currently recommend opioid reduction in bariatric surgery. Both systemic analgesics and regional approaches such as transversus abdominis plane (TAP) block, intraperitoneal and wound modalities, and neuraxial techniques are being used for postoperative pain control in bariatric surgery with some success.

Ultrasound-guided erector spinae plane block is a novel regional anesthesia technique where local anesthetic agent is injected deep into the erector spinae muscle to the fascial plane and allowed to diffuse in caudal and cranial direction. It has been shown effective in a number of conditions such as thoracic surgery/trauma, painful conditions of the limbs, cardiac surgery, breast surgery, and abdominal surgery. To date, only few studies examined the use of ESPB in bariatric surgery, all indicating potential benefits of the technique in terms of opioid sparing and pain control.

This study aimed to compare bilateral ultrasound-guided erector spinalis plane block technique with controls who received bupivacaine injection to the trocar sites, in terms of intraoperative opioid consumption, postoperative pain control in the first 24 hours, and need for rescue analgesic.

METHODS

Patients Sixty-two patients with morbid obesity who underwent laparoscopic bariatric/metabolic surgery (sleeve gastrectomy or gastric bypass) were included in this randomized study.

Patients were required to have a BMI ≥40 kg/m 2 and ASA physical status class 2 or 3.

Exclusion/drop-out criteria were as follows: any complication (allergic reaction or local anesthesia-related complication), failure, or patient refusal during the block procedure; switch to open surgery or a change in the planned surgical protocol; analgesia nociception index (ANI) and/or bispectral index (BIS) monitoring not possible; or patient does not provide consent or withdraws consent at any point after inclusion.

The study protocol was approved by local ethics committee (Ethics Committee for Clinical Studies, Marmara University, Medical Faculty; date, January 3, 2020; number, 09.2020.128).

All patients provided informed consent prior to study entry and the study was conducted in accordance with the Declaration of Helsinki.

Randomization to the study groups Patients were randomly assigned to the erector spina plane block (ESPB) group or the control group using sealed envelopes with 1:1 ratio. ESPB group received ultrasound-guided bupivacaine and lidocaine injection at T9 vertebral level before anesthesia induction. Control group received 5 ml 0.5% bupivacaine injection to each trocar site (total of 25 ml) at the beginning of the operation.

Erector spinalis plane block technique

An experienced anesthesiologist performed ESPB in all patients in sitting position bilaterally.

A linear ultrasound probe (6-13 MHz) was used for ultrasound guidance. Injection was done using in-plane technique. A 22G block needle (100mm, B-Braun, Germany) was inserted 3- cm lateral to the T9 spinous process and advanced in cranio-caudal direction. To separate erector spina muscle from the transverse process, initially 1-2 ml saline was injected; then 20ml 0.5% bupivacaine and 5 ml 0.2% lidocaine were injected following separation. Diffusion of the drugs in erector spina plane at cranio-caudal line was ensured. No analgesic or sedative was used during the procedure.

Intraoperative anesthesia management Anesthesia was induced with propofol 2.5-3.5 mg/kg and 1 mcg/kg bolus dose of remifentanil, which was followed by rocuronium 0.6 mg/kg to aid intubation. Corrected body weight (CBW) was used for the dose adjustment of propofol, and ideal body weight (IBW) was used for the dose adjustments of remifentanil and rocuronium. Total intravenous anesthesia with propofol and remifentanil was used for maintenance and the initial doses were as follows: propofol 6-10 mg/kg/h and remifentanil 0.5 mcg/kg/h. Propofol and remifentanil dose was adjusted to keep BIS between 40 and 45, and ANI between 50 and 70, respectively. Electrocardiography, non-invasive blood pressure, bispectral index (BIS, Medtronic, Mineapolis), and ANI were continuously monitored and recorded at every 30 minutes.

To evaluate perioperative pain and to adjust opioid dose, ANI was continuously monitored throughout the surgical procedure. Two ANI electrodes were placed on the sternum and at the level of left nipple (to the same places with V1 and V5 ECG electrodes, respectively). Total remifentanil dose was recorded for each patient. Depth of anesthesia was monitored to adjust propofol dose using BIS (Aspect Medical Systems, Natick, Mass, ABD).

Fifteen minutes before the completion of the surgical procedure, both groups received 1 g paracetamol and the control group received 150 mg tramadol.

Assessments The primary outcome measure was total intraoperative opioid consumption, and the secondary outcome measure was the change in postoperative pain as assessed by 10-point visual analogue scale (VAS). A blinded investigator recorded self-assessed VAS scores of the patients upon awakening and at 6, 12, and 24 hours. In case VAS ≥ 4, rescue analgesic was given (100 mg tramadol). Timing of first analgesic requirement was recorded.

Statistical analysis Data were analyzed using SPSS (Statistical Package for Social Sciences) version 21 software. Mean ± standard deviation or median (range) was used to express descriptive data. Both hypothesis tests and graphical method were used to test the distribution of continuous variables. Student t test for independent samples or Mann-Whitney U test was used to test between-group differences. Fisher's exact test was used to compare the two groups in terms of complication frequencies. Two-way ANOVA test for repeated measurements was used to examine the significance of differences between groups in postoperative VAS scores and intraoperative measurements over time. Two-sided p values <0.05 were considered indication of statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Patients were required to have a BMI ≥40 kg/m
* ASA physical status class 2 or 3.

Exclusion Criteria:

* any complication (allergic reaction or local anesthesia-related complication)
* failure, or patient refusal during the block procedure
* switch to open surgery or a change in the planned surgical protocol
* analgesia nociception index (ANI) and/or bispectral index (BIS) monitoring not possible
* patient does not provide consent or withdraws consent at any point after inclusion.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-01-03 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
total intraoperative opioid consumption, | postoperatif first 24 hours
  To evaluate intraoperatif opioid consumption, ANI was continuously monitored throughout the surgical procedure.

SECONDARY OUTCOMES:
measure vas the change in postoperative pain | up to 6, 12, and 24 hours.
  measure vas the change in postoperative pain as assessed by 10-point visual analogue scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: MELIHA ORHON ERGUN, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No